CLINICAL TRIAL: NCT00124644
Title: A Phase I Study of R115777 (Zarnestra) in Combination With Induction Chemotherapy in Patients With Newly Diagnosed, High Risk Acute Myeloid Leukemia
Brief Title: Combination Chemotherapy and Tipifarnib in Treating Patients With Newly Diagnosed Acute Myeloid Leukemia
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Withdrawn due to "toxicity" problems
Sponsor: Ohio State University Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000437105; OSU-05020; OSU-2005C0024; NCI-6623
Record Dates: First submitted 2005-07-26; First posted 2005-07-28 (Estimated); Last update posted 2013-05-03 (Estimated); Status verified 2008-01

CONDITIONS: Leukemia
Keywords: adult acute myeloid leukemia with 11q23 (MLL) abnormalities; adult acute myeloid leukemia with t(16;16)(p13;q22); untreated adult acute myeloid leukemia; secondary acute myeloid leukemia
MeSH Terms: conditions — Leukemia; Congenital Abnormalities | interventions — Cytarabine; Daunorubicin; Etoposide; tipifarnib; Drug Therapy

INTERVENTIONS:
Drug: cytarabine
Drug: daunorubicin hydrochloride
Drug: etoposide
Drug: tipifarnib
Procedure: chemotherapy
Procedure: enzyme inhibitor therapy
Procedure: high-dose chemotherapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as cytarabine, daunorubicin, and etoposide, work in different ways to stop the growth of cancer cells, either by killing the cells or by stopping them from dividing. Tipifarnib may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth. Giving combination chemotherapy together with tipifarnib may kill more cancer cells.

PURPOSE: This phase I trial is studying the side effects and best dose of tipifarnib when given together with combination chemotherapy in treating patients with newly diagnosed acute myeloid leukemia.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the maximum tolerated dose of tipifarnib when given in combination with induction therapy comprising cytarabine, daunorubicin, and etoposide followed by consolidation therapy comprising high-dose cytarabine in patients with newly diagnosed high-risk acute myeloid leukemia.

Secondary

* Determine the qualitative and quantitative toxic effects of this regimen, in terms of organ specificity, time course, predictability, and reversibility, in these patients.
* Determine the rate of complete remission in patients treated with this regimen.
* Determine the remission duration, overall survival, and relapse-free and event-free survival of patients treated with this regimen.
* Determine the pharmacokinetics of this regimen in these patients.
* Correlate pharmacodynamic measurements and levels of tumor necrosis factor-alpha with clinical response in patients treated with this regimen.

OUTLINE: This is a dose-escalation study of tipifarnib.

* Induction therapy: Patients receive cytarabine IV continuously on days 1-7; daunorubicin IV and etoposide IV over 2 hours on days 5-7; and oral tipifarnib twice daily on days 5-12.

Patients undergo bone marrow biopsy on day 17 OR days 17 and 24 (if day 17 bone marrow biopsy shows suspicious disease). Patients achieving a complete remission (CR) proceed to consolidation therapy. Patients with residual disease, defined as > 5% leukemic blasts in a bone marrow of ≥ 20% cellularity, receive a second course of induction therapy comprising cytarabine IV continuously on days 1-5; daunorubicin IV and etoposide IV over 2 hours on days 4 and 5; and oral tipifarnib twice daily on days 4-9. Patients achieving a CR after a second course of induction therapy proceed to consolidation therapy. Patients not achieving a CR after a second course of induction therapy are removed from the study.

Cohorts of 3-6 patients receive escalating doses of tipifarnib until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity. An additional 12 patients are treated at the MTD.

* Consolidation therapy: Patients receive high-dose cytarabine IV twice daily on days 1, 3, and 5. Treatment repeats approximately every 6-8 weeks for 4 courses.

After completion of study treatment, patients are followed every 3-6 months for up to 5 years.

PROJECTED ACCRUAL: A maximum of 30 patients will be accrued for this study within 10-15 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed acute myeloid leukemia (AML) according to the WHO classification system

  * High-risk disease
  * Newly diagnosed disease
  * Patients with secondary AML due to prior chemotherapy for a different malignancy are eligible
* No known inv(16), t(8;21), or t(15;17) cytogenetic abnormality
* No acute promyelocytic leukemia
* No CNS leukemia

PATIENT CHARACTERISTICS:

Age

* 18 to 59

Performance status

* ECOG 0-2

Life expectancy

* More than 6 months

Hematopoietic

* Not specified

Hepatic

* AST and ALT ≤ 2.5 times upper limit of normal
* Bilirubin normal

Renal

* Creatinine normal OR
* Creatinine clearance ≥ 60 mL/min

Cardiovascular

* Ejection fraction > 50% by echocardiogram or MUGA
* No symptomatic congestive heart failure
* No unstable angina pectoris
* No cardiac arrhythmia

Immunologic

* No known HIV positivity
* No history of allergic reactions attributed to compounds of similar chemical or biological composition to tipifarnib
* No allergy to imidazoles (e.g., clotrimazole, ketoconazole, miconazole, or econazole)
* No ongoing or active infection

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No other uncontrolled illness
* No psychiatric illness or social situation that would preclude study compliance

PRIOR CONCURRENT THERAPY:

Biologic therapy

* No concurrent epoetin alfa

Chemotherapy

* See Disease Characteristics
* No prior chemotherapy for AML or myelodysplastic syndromes except hydroxyurea

Endocrine therapy

* Not specified

Radiotherapy

* No concurrent palliative radiotherapy

Surgery

* Not specified

Other

* More than 30 days since prior investigational agents
* No other concurrent investigational or commercial agents or therapies for the malignancy

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30
Dates: Start 2006-03; Primary Completion 2007-12 (Actual); Study Completion 2008-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William G. Blum, MD, Principal Investigator — Ohio State University Comprehensive Cancer Center
Locations (1):
- Arthur G. James Cancer Hospital and Solove Research Institute at Ohio State University Medical Center, Columbus, Ohio, United States